CLINICAL TRIAL: NCT06081725
Title: Playfulness in Online and Face-to-face Interactions, From Adulthood to Aging: Physiological, Cognitive, and Emotional Mechanisms and Outcomes
Brief Title: Playfulness in Online and Face-to-face Interactions, From Adulthood to Aging
Acronym: Play
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Shoshi Keisari, Principle Investigator, University of Haifa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 181/22
Record Dates: First submitted 2023-09-29; First posted 2023-10-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Aging; Cognitive Function 1, Social; Social Behavior; Aging Well; Executive Function
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to four arms. At first they will randomly assign to one of two conditions (online or face to face).
  On the second and third session the participants will be randomly assigned to a playful or control interaction.
  The interactions will be separated in a week. A random half of the participants will be assigned to practice the playful interaction at the first week and control interaction in the second week, whereas for the other half this order will be reversed.
Who Masked: Outcomes Assessor
Masking Description: One designated experiment assigned each participant randomly to one of the interactions (playful or control), to keep the other experiments blind to the activity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Playful interactions first session in a face-to-face format (Experimental): Playful interactions operationalized by dramatic improvisation techniques based on verbal and non-verbal elements in a face-to-face format. This arm will take part in the playful interactions in a face-to-face format in the first session and in the active control in the second session
  Interventions: Behavioral: An active control condition in a face-to-face format; Behavioral: Playful interactions in a face to face format
- An active control condition first session in a face-to-face format (Active Comparator): An active control condition that involves introductory conversation and movement exercises in a face-to-face format. This arm will take part in the active control in a face-to-face format in the first session and in the playful interaction in the second session
  Interventions: Behavioral: An active control condition in a face-to-face format; Behavioral: Playful interactions in a face to face format
- Playful interactions first session in an online format. (Experimental): Playful interactions are operationalized by dramatic improvisation techniques based on verbal and non-verbal elements in an online format. This arm will take part in the playful interactions in an online format in the first session and the online active control in the second session
  Interventions: Behavioral: Playful interactions in an online format; Behavioral: An active control condition in an online format
- An active control condition first session in an online format (Active Comparator): An active control condition that involves introductory conversation and movement exercises in an online format. This arm will take part in the active control in an online format in the first session and in the online playful interaction in the second session.
  Interventions: Behavioral: Playful interactions in an online format; Behavioral: An active control condition in an online format

INTERVENTIONS:
Behavioral: Playful interactions in an online format — The activity is grounded in dramatic improvisation and comprises several games: a ball game, an association game, a mirror game, a movement story game. The intervention will be conducted by zoom
  Arms: An active control condition first session in an online format; Playful interactions first session in an online format.
Behavioral: An active control condition in a face-to-face format — The activity consisted of three parts: A structured conversation centered around hobbies. In the second part an exercise in words - singular plural. In the third part, participants will be engaged in a movement practice resembling an exercise class.
  Arms: An active control condition first session in a face-to-face format; Playful interactions first session in a face-to-face format
Behavioral: An active control condition in an online format — The activity consisted of three parts: A structured conversation centered around hobbies. In the second part an exercise in words - singular plural. In the third part, participants will be engaged in a movement practice resembling an exercise class. The intervention will be conducted conducted by zoom
  Arms: An active control condition first session in an online format; Playful interactions first session in an online format.
Behavioral: Playful interactions in a face to face format — The activity is grounded in dramatic improvisation and comprises several games: a ball game, an association game, a mirror game, a movement story game.
  Arms: An active control condition first session in a face-to-face format; Playful interactions first session in a face-to-face format

SUMMARY:
Playful interactions have an important role in human sociality. During playful interactions, two individuals continuously co-create an imaginary world together, such as playing roles in an imaginary scene or co-creating synchronized movements together. Playful interactions are characterized by an enhanced sense of flow and joy and have been associated with physical and psychological well-being across the lifespan. This research team and others have shown that playful interactions are particularly beneficial for the older population, which are at higher risk of cognitive decline and social isolation. The overarching aim of this proposal is to conduct an in-depth investigation of the effects of playful interactions, in older population. Specifically the investigators will test the effect of short playful interaction on cognitive measures, as well as social and affective indices, and compare them to a non-playful interaction (such exercise class, or personal conversation).

DETAILED DESCRIPTION:
Play is a crucial activity that supports human beings and animals throughout the life course, and enables individuals to acquire and practice complex physical, cognitive and social and contemplative skills. The term 'play' has many meanings; over the years, psychologists and biologists have tried to define criteria for the identification of playful behavior. Generally speaking, playful behavior is spontaneous and rewarding to the individual, as players play for the sake of playing; it has no immediate utility beside the play itself (as opposed to, for example, rule-governed competitive sports activities). The play occurs outside ordinary reality, yet maintains a relation with it. Playful behavior consists of actions or thoughts, expressed in novel combinations (such as when a parent takes the role of a child); it is grounded in positive social exchanges, in which the individual is more inclined to behave or think in a spontaneous and flexible way.

In the current study, the investigators will focus on a particular form of social playfulness, termed improvised dramatic interactions (IDI), which plays a central role in creative arts therapies and contemplative arts. IDI can occur on different levels, ranging from non-verbal expressions such as emotions, gestures, and postures, to verbal communication, which involve real-time dialogue and narrative progression. It is the act of spontaneous co-creation which requires people to cooperate on a moment-to-moment basis in order to keep playing. The participants continuously exchange, co-adapt, and co-create. Accordingly, IDI is believed to present an ongoing challenge (and provide training) for different aspects of executive functions and to powerfully trigger a multitude of attentional, perceptual, and social processes. Studies of IDI conducted among younger populations point to its tangible beneficial effects on certain aspects of mental health, such as a reduction of depressive and anxiety symptoms and an enhancement of mood and psychological well-being.

Given the potential of IDI to improve mental health, it is surprising that research on this topic is still sparse; frequently, it lacks well matched control activities and underlying mechanisms are not fully understood. In addition, most studies on improvised playful interactions have focused on children, adolescents and young adults. In this study the investigators aim to examine the beneficial effects of a short playful interaction on the cognitive, social, and mood of older people. the investigators will examine changes in indices of mood, mental health, social functioning, cognition compared to an active control intervention. The study also aims to compare between online playful interactions to face to face.

In addition, in the past two decades there has been a shift toward the development of "tailor-made" interventions that fit individual needs and abilities. This trend is especially important in aging, given increased variability in personality and cognitive and sensory characteristics. In the current study, the investigators aim to investigate the mediating role of personality traits and cognitive functions in connection to the beneficial effect of playful interactions in aging.

The investigators hypnotized that playful interactions will induce greater effects on emotional and social indices, as well as on executive functioning, compared to more familiar social interactions. The investigators hypothesize that these effects will be found in older populations. The effects of short-term playful interaction tasks as compared to the matched social control condition will be preserved in the online format. Individuals' characteristics and personality traits will influence the effects of the interaction on the dependent variables.

Participants

80 participants (up to 95, considering attrition).

To detect a significant interaction between conditions and participant groups (ANOVA within-between interactions with repeated measures as a proxy for MLM, with 4 groups, and 6 types of repeated measures), assuming a medium-small effect size (f2 = .20), and a conservative estimate of correlation (r = .33), a sample size of at least 18 in each arm group is required to achieve a power of 0.90, using GPower. The investigators will recruit 20 participants per group expecting attrition.

Procedure

1. The study will take place in six sites including assisted living facilities, community centers and adults day centers in Israel.
2. Participants will be invited by the research assistance to take part in the study.
3. Participants who will be willing to take part in the study will meet with the research team and will read and signed an informed consent form before participating in the study.
4. Following the informed consent signing, base line measures will be collected (traits and cognitive measures) (T0).
5. Following base line assessment participants will be randomly assigned to four arms. At first, they will randomly assign to one of two conditions (online or face to face). The interactions will be separated in a week. A random half of the two conditions of participants (online and face t face) will be assigned to practice the playful interaction at the first week and control interaction in the second week, whereas for the other half this order will be reversed.
6. One designated experiment assigned each participant randomly to one of the two interactions (playful or control), to keep the other experiments blind to the activity.
7. For each participant, separate interactions will be conducted by a different experimenter.
8. These are the four arms:

   * Playful interactions operationalized by dramatic improvisation techniques based on verbal and non-verbal elements in face to face setting
   * Playful interactions operationalized by dramatic improvisation techniques based on verbal and non-verbal elements in online setting
   * An active control condition that involves introductory conversation and movement exercises in face to face setting in face to face setting
   * An active control condition that involves introductory conversation and movement exercises in face to face setting in online setting
9. The interventions will meet the following criteria: a) ease of implementation in an online system; b) a short interaction between 15-20 minutes. Both interactions incorporated bodily movement; however, the playful interaction encompassed elements of co-creation, spontaneity, and innovation, whereas the control interaction adhered to a more conventional and routine approach.
10. The online interactions will take place using the ZOOM video conference software under laboratory conditions.
11. All interactions will be guided by graduate students of the Theatre department at the university of Haifa or drama therapy students or theatre facilitator - the facilitators, who are unfamiliar to the participants. One designated experiment assigned each facilitator randomly to one of the two interactions (playful or control), to keep the other experiments blind to the activity. The facilitators will be randomly assigned to the different interactions, so that for each participants the separate interactions were conducted by a different facilitator.
12. All interactions will be videoed recorded. A fidelity check will be done by the research team every week to make sure each participants was given the correct interaction (playful or control), and that each interaction included all phases in the protocol.
13. Both interactions will commence with a battery of tests and self-reports before (T1) and after each session (T2). The battery of tests was conducted by an experimenter who will be blind to the type of intervention (playful or control).
14. All self-reports and tests will be administered individually in a quiet and well-lighted room before and after each activity. Items will be read aloud to participants when this will be necessary, and responses will be given orally and coded by the researcher. At the end of the initial assessment (T1), participants transitioned to a designated room, equipped with a computer connected to Zoom, or in case of face to face interaction they will meet the facilitator. They will be introduced to the facilitator previously unknown to them and then the experimenter will leave (so they won't be able to know which intervention will be delivered). Each interaction (playful or control) will be administered by a different and unfamiliar experimenter.
15. At the end of the interaction, participants reconvene with the primary researcher for the administration of the second assessment (T2). It is important to note that the investigators will take pains to ensure that the experimenter administering the initial and second assessment will be blind to the experimental condition.

Dependent variables

At base line (T0):

1. Cognitive tests: forward and backward digit span (WISC III, 1991), phonetic fluency taken (Kave, 2005) from the Hebrew version of the WAIS-IV, ANT attention network test (for younger adults), flanker task (for older adults).
2. Traits (openness to experience and extraversion), attachment styles, novelty seeking and social anxiety will be assessed as control variables and for exploratory analysis to investigate sub-populations for whom playful interactions are most beneficial.

Pre interaction (T1)

* Mood Post interaction (T2)
* Cognitive tests
* Mood
* Flow Questionnaire
* Subjective Arousal
* Closeness
* Perceived Partner Responsivness
* Freiburg Mindfulness Inventory

Data analysis

To test the effects of playful interactions in all of the above measures and experiments the investigators use various tools. As the investigators do not wish to assume equality of variance and a normal distribution, they will apply a mixed-level linear model (MLM). The various measures (cognitive, social, and emotional measures) will serve as the dependent variables; age group (young vs. older adults) and platform (online or F2F) as the between-participant variables, and time of testing (before vs. after) and experimental condition (playful interaction vs. control) as the repeated measures. Follow-up analyses will attempt to find connections between the different dependent measures and relate it to the different experimental groups, traits and age groups. This will be done in exploratory mediation and moderation analyses as well as by correlation analysis

ELIGIBILITY:
Inclusion Criteria:

1. Healthy cognitive functioning for this age-range with a Mini-Mental State Examination above 24, as reported by the community centers or adult day centers
2. No history of auditory or visual pathology, as indicated in a self-report
3. No known clinical diagnosis of a major psychiatric disorder or drug/alcohol abuse, as reported by social worker at the community center and self report
4. Speaking Hebrew
5. Participants who will complete the three study sessions
6. Age above 60 years old.

Exclusion Criteria:

1. Mini-Mental State Examination beyond 25, as reported by the community centers or adult day centers
2. Participants whose responses indicate that they did not follow or did not understand instructions
3. Participants with auditory or visual pathology, as indicated in a self-report
4. Participants who do not speak Hebrew.
5. Participants who will not complete the three study sessions

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Digit span | (1) Base line (2) one week following baseline and immediately after the first interaction (3) two weeks following baseline and immediately after the second interaction
  Digit Span test. consists of two stages (WISC III, 1991): a) Forward Digit Span to evaluate short-term memory. b) Backward Digit Span to assess working memory.
Phonetic fluency | (1) Base line (2) one week following baseline and immediately after the first interaction (3) two weeks following baseline and immediately after the second interaction
  Phonetic fluency taken (Kave, 2005) from the Hebrew version of the WAIS-IV,
Flanker task | (1) Base line (2) one week following baseline and immediately after the first interaction (3) two weeks following baseline and immediately after the second interaction
  (Fan et al., 2005, 2009) attention - response time for correct answers
Perceived Partner Responsiveness | (1) Base line (2) one week following baseline and immediately after the first interaction (3) two weeks following baseline and immediately after the second interaction
  Perceived Partner Responsiveness (Reis et al. 2017). A 4-item questionnaire will asses how one partner perceived the other. It will enable us to assess a relationship's development after these short interactions between unfamiliar partners.
Closeness | (1) one week following baseline and immediately after the first interaction (2) two weeks following baseline and immediately after the second interaction
  was measured using a 3-item questionnaire found in Golland et al., 2019). Participants rated the degree to which they felt closeness, similarity and rapport towards the experimenter during the interaction toward the experimenter on a seven-point Likert scale from 1 (strongly disagree) to 5 (strongly agree): "During the experiment, I felt that I became closer to the other participant?".
Mood | (1) Base line (2) one week following baseline, before and immediately after the first interaction (3) two weeks following baseline, before and immediately after the second interaction
  Mood will be assessed on the Positive and Negative Affect Schedule (Watson et al., 2008), a self-report inventory divided into two subscales assessing positive and negative affect. The inventory consists of 10 items for each subscale, scored on a scale ranging from 1 (very slightly or not at all) to 5 (extremely).

SECONDARY OUTCOMES:
Flow | (1) one week following baseline and immediately after the first interaction (2) two weeks following baseline and immediately after the second interaction
  Flow Questionnaire; a 9-item questionnaire (Csikszentmihalyi, 2000) that measures people's perceived state of flow in a specific context. The scale items reflect the nine flow factors. Participants will be asked to rate items such as "I felt like time passed quickly," "I really enjoyed what I was doing" on a seven-point scale, from 1 (strongly disagree) to 7 (strongly agree). For three dimensions of Flow the full subscale was measured: concentration, transformation of time, autotelic characteristic of the experience and control
Mindfulness | (1) one week following baseline and immediately after the first interaction (2) two weeks following baseline and immediately after the second interaction
  Freiburg Mindfulness Inventory (FMI): A useful, valid and reliable questionnaire for measuring experience of mindfulness during the session with subjects without previous experience with contemplative practice [76]. We adapted the questionnaire to the current study. The adapted inventory consists of 8 items such as: "during the session I was open to the experience of the present moment", on a 5-point scale.
Subjective Arousal | (1) Base line (2) one week following baseline, before and immediately after the first interaction (3) two weeks following baseline, before and immediately after the second interaction
  Subjective Arousal with one item will be measured using a 9-point scale

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Beit-horim, Haifa
  - Beit Avraham - Sephardic community, Haifa
  - Uziel community center for the aging population, Ramat Gan
  - Kibutz Givat Brenner, Rehovot

IPD SHARING:
Plan to Share IPD: Yes
On upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after publication
Access Criteria: Upon request.